CLINICAL TRIAL: NCT01359228
Title: Rifaximin Treatment of Papulopustular Rosacea: Double- Blinded, Placebo-Controlled, Crossover Study
Brief Title: Rifaximin Treatment of Papulopustular Rosacea
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Salix Rifaximin Study
Record Dates: First submitted 2011-04-01; First posted 2011-05-24 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Rosacea
Keywords: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifaximin (Experimental): rifaximin (XIFAXAN®) 1650 mg/day (550 mg tablet three times a day) for 14 days
  Interventions: Drug: Rifaximin (XIFAXAN)
- sugar pill (Placebo Comparator): Placebo 1 tablet three times a day for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin (XIFAXAN) — Rifaximin (XIFAXAN®) 1650 mg/day (550 mg tablet three times a day) for 14 days
  Other Names: XIFAXAN
  Arms: Rifaximin
Drug: Placebo — Placebo 1 tablet three times a day for 14 days.
  Arms: sugar pill

SUMMARY:
The purpose of this study is to determine the effects of rifaximin on skin symptoms in patients with rosacea by double-blinded, placebo-controlled, crossover study.

DETAILED DESCRIPTION:
100 patients will be randomized into two groups.

Group A will receive one rifaximin 550 mg tablet three times a day (1650 mg/day) for 14 days, and after a 4-week washout period, receive one placebo tablet three times a day for 14 days.

Group B will receive placebo first, and then rifaximin with the same dosage schedule to Group A.

Assessments will be performed before application and 4 weeks after the last dosage, for both of rifaximin and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* > 18 years of age with rosacea defined as:
* 3-40 papules/pustules and < 2 nodules,
* A score of 2-4 on the Investigator Global Assessment

Exclusion Criteria:

* Untreated pancreatic insufficiency
* Crohn's disease
* Ulcerative colitis
* Active celiac disease by clinical history
* End stage renal failure
* Less than 18 years old
* Pregnancy or positive pregnancy test
* Rosacea subtype 1 (no papules )
* Topical or oral antibiotics within 4 weeks
* Acne treatments within 4 weeks prior to randomization
* Systemic retinoids within 90 days
* Topical or systemic corticosteroids 4 weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Investigator's Global Assessment (IGA) Score of Rosacea Symptoms | 14 days
  A response to treatment is defined as the achievement of an IGA score of '0 or 1' at endpoint for moderate to severe patients and achievement of an IGA score of '0' at endpoint for mild patients.

SECONDARY OUTCOMES:
Achieving an IGA score of 0. | 14 days
  Percentage of patients achieving an IGA score of '0' (cleared).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Steinhoff, MD, Ph.D., Principal Investigator — UCSF, Dept. of Dermatology
Locations (1):
- UCSF, CTSI, 12-Moffitt/Long Hospital, San Francisco, California, United States